CLINICAL TRIAL: NCT01472718
Title: Efficacy of Thromboaspiration in Patients With High Thrombotic Burden Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Thromboaspiration in Patients With High Thrombotic Burden Undergoing Primary Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Prof. Anna Sonia Petronio, Head of Cardiac Catheterization Laboratory, University of Pisa, Azienda Ospedaliero-Universitaria Pisana, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP-DCT-201001
Record Dates: First submitted 2011-11-13; First posted 2011-11-16 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Primary PCI for STEMI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard primary coronary intervention (Active Comparator)
  Interventions: Device: standard primary PCI (with stenting, as required)
- coronary thrombectomy (Experimental)
  Interventions: Device: coronary thrombectomy

INTERVENTIONS:
Device: coronary thrombectomy — coronary thrombectomy with either Angiojet device (rhelytic thrombectomy) or Export device (manual aspiration)
  Arms: coronary thrombectomy
Device: standard primary PCI (with stenting, as required) — standard primary PCI (usually with stenting) for STEMI, without use of thrombectomy or distal protection devices
  Arms: standard primary coronary intervention

SUMMARY:
200 consecutive patients presenting with STEMI within 12 hours from the onset of symptoms and having a high thrombotic burden at coronary angiography, defined as the presence of a thrombus size ≥ 2 times the diameter of the vessel, according to a visual estimate. The main objective of the study is to evaluate the effectiveness of thrombectomy (either rheolytic or manual aspiration) as an adjunct to primary or rescue angioplasty, in patients with angiographic evidence high thrombotic burden in the culprit artery. Primary end points: (1) rate of complete ST-segment elevation resolution at 60 minutes after the end of the procedure; (2) infarct size as assessed by delayed-enhancement cardiac magnetic resonance imaging (DE-MRI) at 3 months after the index procedure.

Secondary endpoints: post-procedural TIMI flow grade; post-procedural MBG; infarct transmurality at 3 months; MVO at 3 months; 1-year actuarial freedom from MACEs.

ELIGIBILITY:
Inclusion Criteria:

1. Prolonged, continuous signs and symptoms of ischemia lasting more than 20 min, starting within 12 hours prior to randomization, and ST elevation ≥ 2mm in ≥2 contiguous ECG leads, or new left bundle branch block (LBBB)
2. Presence of high thrombotic burden in the culprit lesion at diagnostic angiography (defined as the presence of a thrombus size ≥ 2 times the diameter of the vessel, according to a visual estimate, or abrupt cut-off occlusion of a coronary artery ≥3 mm in reference vessel diameter)
3. Written informed consent

Exclusion Criteria:

* Low-risk (ST elevation in ≤2 leads) inferior AMI
* Previous infarction in the same area (assessed by ECG)
* PCI in the 2 weeks prior to AMI
* Active internal bleeding
* History of cerebrovascular accident in the previous 2 years or cerebrovascular accident with a significant residual neurological deficit
* Head or spine surgery or trauma in the previous 2 months
* Recent (within six weeks) gastrointestinal (GI) or genitourinary (GU) bleeding of clinical significance
* Administration of oral anticoagulants within seven days unless prothrombin time is <1.2 times control
* Bleeding diathesis or severe uncontrolled arterial hypertension
* Thrombocytopenia (<100 000 cells/mL)
* Recent (within six weeks) major surgery or trauma
* Intracranial neoplasm, arteriovenous malformation, or aneurysm
* Severe renal or liver failure
* Allergy to aspirin
* Contraindication to MRI examination
* Pregnancy and lactation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

REFERENCES:
- [Derived] De Carlo M, Aquaro GD, Palmieri C, Guerra E, Misuraca L, Giannini C, Lombardi M, Berti S, Petronio AS. A prospective randomized trial of thrombectomy versus no thrombectomy in patients with ST-segment elevation myocardial infarction and thrombus-rich lesions: MUSTELA (MUltidevice Thrombectomy in Acute ST-Segment ELevation Acute Myocardial Infarction) trial. JACC Cardiovasc Interv. 2012 Dec;5(12):1223-30. doi: 10.1016/j.jcin.2012.08.013. PMID 23257370

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Primary Coronary Intervention | Coronary Thrombectomy
Started | 104 | 104
Completed | 98 | 97
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Primary Coronary Intervention | Coronary Thrombectomy | Total
Number analyzed (Participants) | 104 | 104 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 58 | 118
  >=65 years | 44 | 46 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [54 to 70] | 63 [53 to 71] | 62 [53 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 16 | 41
  Male | 79 | 88 | 167
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 104 | 104 | 208
coronary TIMI frame count [Mean (Standard Deviation); unit: frames] | 86 (28) | 95 (17) | 91 (25)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete ST-segment Elevation Resolution at 60 Minutes After the End of the Procedure
Time Frame: 60 minutes after the end of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Primary Coronary Intervention | Coronary Thrombectomy
Number analyzed (Participants) | 104 | 104
Participants | 38 | 58

2. Primary Outcome: Infarct Size as Assessed by Delayed-enhancement Cardiac Magnetic Resonance Imaging (DE-MRI)
Time Frame: 3 months after the index procedure
Measure: Mean (Standard Deviation); unit: % of LV mass
Arm/Group | Standard Primary Coronary Intervention | Coronary Thrombectomy
Number analyzed (Participants) | 75 | 79
% of LV mass | 19.3 (10.6) | 20.4 (10.5)

ADVERSE EVENTS:
Arm/Group | Standard Primary Coronary Intervention | Coronary Thrombectomy
All-Cause Mortality (participants affected / at risk) | 2/104 | 2/104
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/104
Other Adverse Events (participants affected / at risk) | 0/104 | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No